CLINICAL TRIAL: NCT02396615
Title: SATIN WP4 - The Acute Effect on Appetite of Pineapple Juice With Viscofiber and Red Ginseng
Brief Title: SATIN WP4 Acute Effect on Appetite of Pineapple Juice With Viscofiber and Red Ginseng
Acronym: SATIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University of Leeds (Other); University of Liverpool (Other)
Responsible Party: Principal Investigator, Anders Mikael Sjödin, MD, PHD ass professor, Dr, PhD, Associate Professor,, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: B318
Record Dates: First submitted 2015-02-19; First posted 2015-03-24 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: Ad libitum energy intake; Appetite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): Satin pineapple. Active juice with fibre and ginseng
  Interventions: Dietary Supplement: SATIN pineapple
- Control (Placebo Comparator): SATIN pineapple control. Control juice - normal juice prpoducts without added active ingredients
  Interventions: Dietary Supplement: SATIN pineapple control

INTERVENTIONS:
Dietary Supplement: SATIN pineapple — Active juice with added fibre and ginseng
  Arms: Active
Dietary Supplement: SATIN pineapple control — Control products without active ingredients
  Arms: Control

SUMMARY:
The objective of the study is to establish whether a Pineapple juice with Viscofiber and Red ginseng can enhance satiety and reduce appetite and/or accelerate satiation in the short-term.

DETAILED DESCRIPTION:
A double-blind, randomised crossover design will be employed with an experimental (active) condition and a control condition at least one week apart. After having successfully completed screening procedures eligible participants will be invited for two separate test days, at least 7 days apart. On the two test days, the products will be provided in a randomized order as part of a fixed breakfast meal, and subjective appetite ratings will be measured every 30 min for the following 8 hours. Satiety and satiation will be measured through administration of test meals in the laboratory supplied with controlled food intake under free-living conditions

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided written informed consent
* Healthy men and women
* Ages between 18 and 55 years
* BMI between 25.0-31.9 kg/m2
* Regular breakfast eaters (eating breakfast ≥ 4 times a week)
* Regular menstrual periods (women only)

Exclusion Criteria:

* Significant health problems as judged by the investigator
* Taking any medication or supplements known to affect appetite or body weight within the past month and/or during the study as judged by the investigator
* Pregnant, planning to become pregnant within the next 4 weeks or breastfeeding (women only)
* History of anaphylaxis to food
* Any known food allergies or food intolerance
* Smoking, smoking cessation within the past 3 months or nicotine use (electronic cigarettes)
* Self-reporting currently dieting or having lost/gained significant amount of weight (±3 kg) in the previous 3 months
* Significant changes in physical activity patterns in the past 4 weeks or intention to change during the study as judged by the investigator
* Significant change in diet in the past 4 weeks or intention to change the diet during the study as judged by the investigator
* Use of systemic or local treatment likely to interfere with evaluation of the study parameters as judged by the investigator
* Participants who work in appetite or feeding related areas
* Participants not able to comply with the study protocol
* Post-menopausal (women only)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Ad libitum energy intake | Baseline (week 0)
  Total ad libitum energy intake during test day 1
Ad libitum energy intake | Test day 2 (week 1)
  Total ad libitum energy intake during test day 2

SECONDARY OUTCOMES:
VAS score for appetite sensation - hunger | Every 30 min during test day 1 and test day 2
  Perceptions of hunger, assessed using 100 mm VAS scales
Eating behaviour questionnaire - binge eating scale | Screening
  Questionnaire by Gormally et al. 1982
Eating behaviour questionnaire - Control of Eating | screening
  Questionnaire by Hill et al. 1991
Eating behaviour questionnaire - three factor eating questionnaire | screening
  Three Factor Eating Questionnaire by Stunkard and Messick, 1985
Eating behaviour questionnaire- power of food | screening
  Power of food scale by Lowe et al 2009
VAS score for appetite sensation - fullness | every 30 min during test day 1 and test day 2
  Perceptions of fullness, assessed using 100 mm VAS scales
VAS score for appetite sensation - Desire to eat | every 30 min during test day 1 and test day 2
  Perceptions of Desire to eat, assessed using 100 mm VAS scales
VAS score for appetite sensation - prospective consumption | every 30 min during test day 1 and test day 2
  Perceptions of prospective suncumption, assessed using 100 mm VAS scales

CONTACTS AND LOCATIONS:
Overall Officials: Anders Sjödin, Dr, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Frederiksberg, Denmark